CLINICAL TRIAL: NCT05701943
Title: Home- vs Gym-based Exercise Delivery Modes of Two Aerobic Training Regimes on Cardiorespiratory Fitness and Arterial Stiffness in Adults With Intellectual and Developmental Disability During the COVID-19 Pandemic
Brief Title: Comparison of Home- vs. Gym-based Exercise Delivery Modes
Acronym: UPSIDE DOWNS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Collaborators: Ginásio Clube Português (Unknown); Faculdade de Motricidade Humana - Universidade de Lisboa (Unknown); Universidade Europeia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UPSIDE DOWNS
Record Dates: First submitted 2023-01-04; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Vascular Stiffness; Cardiorespiratory Fitness
Keywords: Covid-19; Pulse wave velocity; Cardiovascular disease; Physical exercise
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases; Motor Activity | interventions — Home Care Services, Hospital-Based

STUDY DESIGN:
Intervention Model Description: This study was a randomized controlled trial, where a convenience group of 17 were randomized in a 1:1 ratio to an SIT or CAET regime by using a random-block randomization scheme. Participants in both aerobic regimes received a 16-week supervised exercise program performed 3 times a week for 60 min each session. The intervention started with 8 weeks of online training via Google Meets at their homes followed by 1 month of detraining with no exercise sessions besides those made available by the SPORTS4ALL program, and another 8 weeks of on-site training at the gym. During the intervention, adherence to the protocols were assessed with an exercise diary. Schedule of enrolment, intervention, and assessments for the duration of the study are displayed in Supplement 1. Assessments were conducted on 4 occasions over a 20-week period: before (M1; 0 weeks) and after (M2; 8 weeks) the home-based intervention; and before (M3, 12 weeks) and after (M4; 20 weeks) the gym-based intervention.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sprint Interval Training (Experimental): The SIT consisted of a combination of aerobic, resistance, balance, and flexibility exercises. Exercise started with 5 min of warm-up followed by bouts of 5-10 min of exercise consisting of 5-20 s all-out sprints followed by 15-45 s of low cadence recovery (1:3-1:2 work-rest ratio). The duration of the sprints and active recovery were modified throughout the program. To ensure that participants exercised at the appropriate intensity, the OMNI scale 8-10 (Stanish & Aucoin, 2007) was applied during the home intervention, and an HR chest band (H10 Polar, Electro, Kempele, Finland) was used during the gym intervention.
  Interventions: Behavioral: Home-Based; Behavioral: Gym-Based
- Continuous Aerobic Exercise Training (Active Comparator): CAET was based on a combination of aerobic, resistance, balance, and flexibility exercises. The exercise on the cycle ergometer started with 5-min of warm-up followed by 3 bouts of continuous cycling at a steady-state intensity. The duration of the bouts (5-10 min) and the intensity (55-85% HRR) were progressively increased throughout each phase. To ensure that the participants exercised at the appropriate intensity, the OMNI scale 4-6 (Stanish & Aucoin, 2007) was used during the home-based intervention, and an HR chest band (H10 Polar, Electro, Kempele, Finland) was worn during the gym-based intervention.
  Interventions: Behavioral: Home-Based; Behavioral: Gym-Based

INTERVENTIONS:
Behavioral: Home-Based — During the home-based intervention, aerobic training was performed using body weight exercises such as jumping jacks, standing box, side shift with floor touch, high knees, half burpee, and hook box (Borrega-Mouquinho et al., 2021).
Behavioral: Gym-Based — During the gym-based intervention, aerobic training was performed on cycle ergometers (Star Trac Spinner Blade ION 7220, Vancouver, WA).

SUMMARY:
Home-based exercise interventions were the only alternatives to attenuate physical deconditioning and ameliorate traditional and emergent cardiovascular risk factors progression during the COVID-19 outbreak. Benefits in physical and psychological health have only been reported in adults without intellectual and developmental disability (IDD).

The purpose of this study is to compare home vs gym-based delivery exercise modes of two 8-week supervised aerobic training regimes on cardiorespiratory fitness and arterial structure and stiffness in adults with IDD.

It is hypothesized that home- and gym- based exercise delivery modes will be equally effective in improving cardiorespiratory fitness and overall arterial heath, although in an intensity dependent manner. A secondary analysis examining changes in blood pressure and body composition will be performed.

DETAILED DESCRIPTION:
A total of 40 participants from the project SPORTS4ALL by Ginásio Clube Português (GCP) were recruited to participate in the study. Study advertising took take place through direct invitation by the research team and rehabilitation technicians. The time frame for recruitment of participants take approximately 1 month. Eligible volunteers were invited to an initial meeting with their families/legal guardians, exercise physiologists, and rehabilitation technicians. During this meeting, the procedures of the trial, testing procedures, benefits, risks, and the time required for the study will be explained. In addition, an information sheet about the research and an informed consent form for participants and parent(s)/ legal guardian(s), in accordance with the approval by the Ethical Committee of Faculdade de Motricidade Humana - Universidade de Lisboa, was distributed. Informed written consent were signed by participants and parent(s) legal guardian(s) before allocation. After signing the informed consent, participants or parents/legal guardians were asked to answer the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) questionnaire, to assess their readiness to increase their levels of physical activity, and a sociodemographic data questionnaire. During a second visit, all volunteers participated in familiarization sessions before baseline testing at the laboratory. The number of familiarization sessions was repeated until the researchers observed that the participants are confident and able to perform all assessments correctly (1-2 sessions). Of the 36 participants recruited, by the time the mandatory COVID-19 home confinement was declared by the Portuguese government, only 17 participants had completed laboratorial exercise testing. Only these participants were part of the present study.

This study was a randomized controlled trial, where a convenience group of 17 who had completed laboratory exercise tests, were randomized in a 1:1 ratio to an SIT or CAET regime by using a random-block randomization scheme. Participants in both aerobic regimes received a 16-week supervised exercise program performed 3 times a week for 60 min each session. The intervention started with 8 weeks of online training via Google Meets at their homes followed by 1 month of detraining with no exercise sessions besides those made available by the SPORTS4ALL program, and another 8 weeks of on-site training at the gym. During the intervention, adherence to the protocols were assessed with an exercise diary. Assessments were conducted on 4 occasions over a 20-week period: before (M1; 0 weeks) and after (M2; 8 weeks) the home-based intervention; and before (M3; 12 weeks) and after (M4; 20 weeks) the gym-based intervention. During M1, assessments and personal information was obtained. All laboratory tests were conducted by the same researchers during the morning. Participants were asked to refrain from eating for at least 3 h, alcohol for 24 h, caffeine for 8 h, and vigorous exercise for 48 h before data collection. All laboratorial evaluations were performed on a single day of testing at each measurement round. On this day, the participants had their (1) body composition measured and then quietly rest for at least 15 min in the supine position before data collection in the following order: (2) brachial arterial pressure, (3) carotid intima media thickness, (4) stiffness indices by carotid vascular ultrasound, (5) regional arterial stiffness by applanation tonometry and (6) an incremental test to exhaustion.

The exercise regimes were delivered at participants' homes for 8 weeks via Google Meets and at the gym during an identical period. All sessions were designed by experienced exercise physiologists together with rehabilitation technicians, following the guidelines of the American College of Sports Medicine (ACSM) and the National Strength and Conditioning Association (NSCA). Exercise physiologists in charge of delivering the interventions underwent standardized training to ensure that the sessions offered were comparable and went through a 2-month familiarization period where they observed the exercise sessions from the project SPORTS4ALL by GCP, met the participants, and led exercise activities, while under the supervision of the responsible Rehabilitation Technicians of the project SPORTS4ALL. During this period, the rating of perceived exertion was reinforced using the OMNI scale. The multi-component exercise programs included aerobic, resistance, balance, and flexibility training. Both SIT and CAET regimes were divided into 2 groups: 8-9 participants/group and the participant-Exercise Physiologist ratio of 3:1, partnered with at least 1 Rehabilitation Technician in each exercise session. Both programs were divided into 3 phases: initial phase (week 1-3); improvement phase (week 4-6); and maintenance phase (week 7-8). Sessions for both regimes were also matched for total duration. All sessions included 5 min of standardized warm-up and cool-down exercises. The warm-up was implemented to gradually increase the HR, body temperature, joint mobility and prepare the body of the participants to the exercises of the conditioning phase. After the conditioning phase, cool-down exercises were performed followed by stretching exercises. During the washout period (4 weeks), 14 participants performed 3 sessions representing each phase of the home-based intervention wearing heart rate monitors to obtain a proxy of the exercise intensity in each phase of the home-based intervention. Resistance training included a total of six exercises: 3 for the upper limbs (seated biceps curl, triceps extension, and frontal shoulder raise); 2 for the torso (1 for the back: seated row and 1 for the abdominals: side bend); and 1 for the lower limbs (chair squats). All exercises were performed with 2-4 kg dumbbells, or the participants' body weight. The intensity of the strength training was monitored using the 0-10 points Rate of Perceived Exertion OMNI- Resistance Exercise Scale (RPE OMNI-RES) validated for resistance training. The intensity of resistance training was kept constant at 2 x 12 rep at RPE OMNI-RES 8, throughout the study period. Balance training was designed to challenge the central and peripheral mechanisms involved in the control of movement and stability (vestibular; visual and somatosensory). Flexibility exercises were performed after the cool-down period of each session. Sustained stretches were used for each major muscle group targeted during the session. Active and passive static stretching exercises were used, holding the position for 10-30 s at a point of tightness or slight discomfort.

Statistical Analyses An intention-to-treat analysis was performed using all randomized participants. The data are presented as mean and standard deviation. The Shapiro-Wilk and Levene tests, as well as plot inspection, were used to verify normality and homoscedasticity assumptions, respectively. To compare baseline individual characteristics independent-samples t-tests were used.

The changes in the cardiorespiratory fitness and vascular outcomes were examined using linear mixed models fitted with restricted maximum likelihood and applying Satterthwaite's method for approximating degrees of freedom for the F test from the R lmerTest package. The fixed effects were time and aerobic regime, whereas the random intercept was defined for each participant. Using the R sjstats package, partial eta squares (η2) were calculated for each main effect and interaction and interpreted as small (η2 < 0.05), medium (η2 < 0.25), and large (η2 > 0.25) effect sizes. In the presence of significant differences in main effects and interactions, post-hoc comparisons using Tukey's HSD test were performed using the R emmeans package. All statistical analyzes were performed with a significant level (α) of < 0.05 using the R software, version 4.1.2.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years and ≤ 55 years
* diagnosed with mild to moderate IDD
* exercised at least 1 d/wk in the last 2 months
* able to participate on group exercise activities with ≥ 8 people
* able to walk independently
* and able to understand and perform all physical fitness assessments.

Exclusion Criteria:

* any form of cardiovascular disease
* significant respiratory disorder
* metabolic disease
* atlanto-axial instability
* severe or profound IDD
* smoking
* and/or use of heart rate (HR) and blood pressure altering or non-steroidal anti-inflammatory medications
* inability to comply with guidelines for participation in exercise testing and training.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness | Assessments were conducted on 4 occasions over a 20-week period: before (M1; 0 weeks) and after (M2; 8 weeks) the home-based intervention; and before (M3, 12 weeks) and after (M4; 20 weeks) the gym-based intervention.
  Each participant performed a ramp incremental cycle ergometer test to exhaustion on a calibrated electronically braked cycle ergometer (Monark 839 E, Ergomedic; Monark, Vansbro, Sweden) at a pedal cadence of 70-75 rev.min-1. The initial and incremental workloads were 10-20 watts. Inspired and expired gases were continuously analyzed, with mixing-chamber gas exchange measurements using a portable gas analyzer (K5, Cosmed, Rome, Italy). Before each test, the O2 and CO2 analyzers were calibrated using ambient air and standard calibration gases of known concentration (16.7% O2 and 5.7% CO2). Heart rate was continuously monitored (Garmin, US) and the participants did not carry the gas analyzer. Data were evaluated in 10 s averages, and peak VO2 (mL/kg/min) was defined as the highest 20-second value attained in the last minute.
Change in Arterial Stiffness | Assessments were conducted on 4 occasions over a 20-week period: before (M1; 0 weeks) and after (M2; 8 weeks) the home-based intervention; and before (M3, 12 weeks) and after (M4; 20 weeks) the gym-based intervention.
  Arterial stiffness as measured by PWV (m/s) from piezoelectric pressure mechanotransducers placed on the carotid, femoral and distal posterior tibial arteries on the right side of the body. The operator positioned the carotid sensor with the help of its specific holder and manually held the femoral sensor on the femoral artery and the distal sensor on the distal posterior tibial artery. The right common carotid artery also was scanned with an Arietta V60 ultrasound machine (Hitachi Aloka Medical Ltd, Mitaka-shi, Japan) using a 7.5-MHz linear array probe incorporating a 5-MHz Doppler transducer. In longitudinal view, the intima of the artery was clearly imaged from both the anterior and posterior walls, and a single scan line was aligned perpendicularly to the vessel walls at a site 20 mm proximal to the carotid bulb. The corresponding displacement waveforms and diameter curve were thus calculated using high-resolution online wall tracking technology, with a sampling rate of 1 kHz.

SECONDARY OUTCOMES:
Change in Arterial Structure | Assessments were conducted on 4 occasions over a 20-week period: before (M1; 0 weeks) and after (M2; 8 weeks) the home-based intervention; and before (M3, 12 weeks) and after (M4; 20 weeks) the gym-based intervention.
  cIMT (mm) measurements were recorded using high-resolution, non-invasive, semi-automated B-Mode ultrasound (Arietta V60; Aloka/Hitachi Medical Systems). The diameter was measured in M-Mode with a high-frequency linear array probe (7.5 MHz). cIMT was measured twice on the far wall of the common carotid artery, 1 cm proximal to the bulb at the end-diastolic moment (R-wave), when cIMT is thickest. The vascular diameter was measured at the same location as cIMT. The average minimum diameter value of the right common carotid artery, which corresponds to end-diastolic cIMT, was recorded from at least 5 heart cycles. Values obtained were compared to estimated age- and sex-specific percentiles of cIMT in populations with different cardiovascular risk profiles.
Change in Body Mass Index | Assessments were conducted on 4 occasions over a 20-week period: before (M1; 0 weeks) and after (M2; 8 weeks) the home-based intervention; and before (M3, 12 weeks) and after (M4; 20 weeks) the gym-based intervention.
  Height (cm) and body weight (kg) were measured to the nearest 0.1 cm and nearest 0.1 kg, respectively, on a scale with an attached stadiometer (model 770, Seca; Hamburg, Deutschland). Body Mass Index (BMI) was calculated as participant's weight in kilograms divided by the square of height (m).
Change in Body Composition | Assessments were conducted on 4 occasions over a 20-week period: before (M1; 0 weeks) and after (M2; 8 weeks) the home-based intervention; and before (M3, 12 weeks) and after (M4; 20 weeks) the gym-based intervention.
  Body composition (%fat; %muscle mass) was measured with a seca mBCA 515 using four pairs of electrodes (eight electrodes in total) positioned in each hand and foot. The 8-electrode technique enables segmental impedance measurement of the arms and legs. By this means, impedance was measured with a current of 100 μA at frequencies between 1 and 1 000 kHz.
Change in Waist Circumference | Assessments were conducted on 4 occasions over a 20-week period: before (M1; 0 weeks) and after (M2; 8 weeks) the home-based intervention; and before (M3, 12 weeks) and after (M4; 20 weeks) the gym-based intervention.
  Waist circumference was measured at the iliac crest (cm) to the nearest 0.1 cm.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Melo, PhD, Principal Investigator — Egas Moniz School of Health and Science
Locations (1):
- Ginásio Clube Português, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in exercise training in intellectual and developmental disability. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact xmelo@egasmoniz.edu.pt.

REFERENCES:
- [Background] Oviedo GR, Guerra-Balic M, Baynard T, Javierre C. Effects of aerobic, resistance and balance training in adults with intellectual disabilities. Res Dev Disabil. 2014 Nov;35(11):2624-34. doi: 10.1016/j.ridd.2014.06.025. Epub 2014 Jul 18. PMID 25041876
- [Background] Oviedo GR, Javierre C, Font-Farre M, Tamulevicius N, Carbo-Carrete M, Figueroa A, Perez-Testor S, Cabedo-Sanroma J, Moss SJ, Masso-Ortigosa N, Guerra-Balic M. Intellectual disability, exercise and aging: the IDEA study: study protocol for a randomized controlled trial. BMC Public Health. 2020 Aug 20;20(1):1266. doi: 10.1186/s12889-020-09353-6. PMID 32819350
- [Background] Borrega-Mouquinho Y, Sanchez-Gomez J, Fuentes-Garcia JP, Collado-Mateo D, Villafaina S. Effects of High-Intensity Interval Training and Moderate-Intensity Training on Stress, Depression, Anxiety, and Resilience in Healthy Adults During Coronavirus Disease 2019 Confinement: A Randomized Controlled Trial. Front Psychol. 2021 Feb 24;12:643069. doi: 10.3389/fpsyg.2021.643069. eCollection 2021. PMID 33716913
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Derived] Melo X, Simao B, Catela C, Oliveira I, Planche S, Louseiro A, Maroco JL, Oviedo GR, Fernhall B, Santa-Clara H. Home- vs gym-based exercise delivery modes of two multicomponent intensity training regimes on cardiorespiratory fitness and arterial stiffness in adults with intellectual and developmental disability during the COVID-19 pandemic - a randomized controlled trial. J Intellect Disabil. 2025 Mar;29(1):66-85. doi: 10.1177/17446295241242507. Epub 2024 Mar 27. PMID 38537027